CLINICAL TRIAL: NCT00933075
Title: Dermatological Evaluation of the Photo Irritation and Photo Sensitivity Potential for Dermacyd Silver Frutal (Lactic Acid).
Brief Title: Dermacyd Silver Frutal (Lactic Acid) - Photo Evaluation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACAC_L_04843
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Hygiene

ARMS (1):
- Dermacyd Silver Frutal (Lactic Acid) (Experimental): Dermacyd Silver Frutal (Lactic Acid) sample will be applied like a curative. Physiologic solution and mineral oil will be also usedas a control sample.
  Interventions: Drug: LACTIC ACID(ND)

INTERVENTIONS:
Drug: LACTIC ACID(ND) — Dermacyd Silver Frutal (Lactic Acid) sample will be applied like a curative for 5 weeks (treatment period).

SUMMARY:
Primary Objective:

To demonstrate the absence of photoirritation and photosensitization potential of the product Dermacyd Silver Frutal.

ELIGIBILITY:
Inclusion criteria:

* Phototype Skin II and III Integral skin test in the region
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion

Exclusion criteria:

* Lactation or pregnancy
* Use of Antiinflammatory 30 days and/or immunossupression drugs for until 3 months before volunteers selection
* Diseases which can cause immunosuppresion, such as diabetes, HIV
* Use of photosensitivity drugs
* History of sensitivity or photosensitivity for topic products
* Cutaneous active disease which can modify the study results
* History or activity of photodermatosis
* Personal or family antecedents of cutaneous neoplasia photo induced
* Presence of injury precursor of cutaneous neoplasia, such as melanociticos nevus and actinic keratosis
* Intense exposure solar in the test region
* Use of new drugs and/or cosmetics during the study
* Previous participation in studies using the same product in test
* Relevant history or confirmation of alcohol or other drugs abuse
* Intolerance detected or suspected for some component of the sample tested
* Medecin or sponsor employees or their close family.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Measure of the photo irritation test and the photosensitivity by using UVA irradiation and evaluation according to International Contact Dermatitis Research Group (ICDRG) scale. Evaluation of the sensibility according to the skin type. | From the treatment start to the end of the study (treatment period 5 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil